CLINICAL TRIAL: NCT02699840
Title: Observational Study of a Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine Menactra® Administered in Individuals 2 Through 55 Years Old Under Standard Health Care Practice in the Russian Federation
Brief Title: Observational Safety Study of Menactra® Administered Under Standard Health Care Practice in the Russian Federation
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: MTA92; U1111-1174-4339 (Other: WHO)
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; Menactra®; Meningococcal Vaccine
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Menactra Study Group 1: Participant aged 2 through 11 years at vaccination
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine
- Menactra Study Group 2: Participant aged 12 through 17 years at vaccination
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine
- Menactra Study Group 3: Participant aged 18 through 55 years at vaccination
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — No vaccine will be provided as part of this study
  Other Names: Menactra®
  Groups: Menactra Study Group 1
Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — No vaccine will be provided as part of this study
  Other Names: Menactra®
  Groups: Menactra Study Group 2
Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — No vaccine will be provided as part of this study
  Other Names: Menactra®
  Groups: Menactra Study Group 3

SUMMARY:
The aim of this study is to generate local data on the safety of Menactra® in individuals 2 to 55 years of age in the Russian Federation.

Primary Objective:

* To describe the safety profile after 1 dose of Menactra® administered in individuals 2-55 years of age under standard health care practices.

DETAILED DESCRIPTION:
Participants will be enrolled after receipt of one dose of Menactra® during a routine health care visit. They will be monitored for safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 through 55 years on the day of enrollment "2 through 55 years" means from the day of the 2nd birthday to the day before the 56th birthday
* For adults (18-55 years old) Informed consent form has been signed and dated by the participant.
* For minors: Informed consent form has been signed and dated by the parent. In addition, in accordance with the Institution Ethics Committee/Institution Review Board requirements and as appropriate for the age of the participant:
* participants aged 14 to 17 years are required to sign and date the informed consent form,
* participants aged 10 to 13 years are required to sign and date the assent form,
* for participants under 10 years, consent may be asked orally according to participant's age and ability for understanding
* Receipt of one dose of Menactra® on the day of inclusion and prior to enrollment into the study, in routine practice according to the approved local product insert.

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the enrollment) or planned participation during the present study period in a clinical study investigating a vaccine, drug, medical device, or medical procedure.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants aged 2 to 55 years will be enrolled after receipt of one dose of Menactra® during a routine health care visit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting solicited injection site and systemic reactions after a single dose of Menactra® vaccine | Day 0 to Day 7 post-vaccination
  Solicited injection site: Pain, Erythema and Swelling, Solicited systemic: Fever (Temperature), Headache, Malaise and Myalgia

SECONDARY OUTCOMES:
Number of participants reporting unsolicited adverse events and serious adverse events after a single dose of Menactra® vaccine | Day 0 to Day 28 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Russia
Locations (1):
- Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com